CLINICAL TRIAL: NCT05919498
Title: Realistic Evaluation of a Job Retention Program After Breast Cancer
Acronym: RECOVA-FTRACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5143
Record Dates: First submitted 2023-02-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; realistic evaluation; investigation; Evaluation of FASTRACS-RCT intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients in the FASTRACS-RCT intervention arm: The individuals in this group are patients in the intervention arm of the FASTRACS-RCT study.
  Once their follow-up for the FASTRACS-RCT study is completed, they will be contacted to participate in the RECOVA-FASTRACS survey. They will be asked to conduct an individual semi-directive interview.
  Patients may agree to provide contact information for people who have accompanied them on their return-to-work journey.
  Interventions: Other: Individual semi-directive interview
- Trajectory persons: Trajectory persons are defined by FASTRACS-RCT patients. These persons have accompanied patients on their return-to-work journey. They may be someone close to you (family, friends, etc.), the general practitioner, a person from the company (colleagues, manager, occupational physician), or other health professionals (nurse, psychologist, etc.).
  As a first step, all trajectory persons will complete an individual semi-directive interview. Then, some will be offered to participate in focus groups
  Interventions: Other: Individual semi-directive interview; Other: Focus groups
- Professionals/Focus group: This group is composed of some of the trajectory persons and professionals who participated in the delivery of the FASTRACS-RCT study intervention tools.
  These individuals will participate in the focus groups.
  Interventions: Other: Focus groups

INTERVENTIONS:
Other: Individual semi-directive interview — This intervention concerns the trajectories of patients who have completed their participation in FASTRACS-RCT. Participant are : patients in the FASTRACS-RCT intervention arm (Groupe 1) and Trajectory persons (groupe 2).
  During the individual interviews, the investigator and the participant will discuss the use of the FASTRACS-RCT tools and the patient's course of care.
  The individual interviews will take place at the location chosen by the participant and will last on average one hour.
  Groups: Patients in the FASTRACS-RCT intervention arm; Trajectory persons
Other: Focus groups — This second intervention will take place at the end of the last patient followed by the FASTRACS-RCT.
  During the focus groups, participants will discuss the use of the FASTRACS-RCT tools.
  The focus groups will take place in a meeting room made available for the occasion and will last on average two hours.
  Groups: Professionals/Focus group; Trajectory persons

SUMMARY:
Returning to and maintaining employment after cancer is essential for restoring social participation, financial independence and reducing the social costs associated with cancer. Many obstacles that prevent or delay the return to work have been identified. They are associated with the consequences of the disease and treatments such as fatigue, pain and cognitive disorders, the lack of collaboration between health professionals (oncologists, general practitioners and occupational physicians), and the characteristics of the environment. in terms of the demands of the job, and the (lack of) social support from superiors and colleagues. There are social inequalities in the return to work after cancer, with a poorer professional prognosis among older and less qualified people. Social inequalities linked to ethnicity have been documented in other countries.

In France, 58,500 new cases of breast cancer are diagnosed each year, half of them in women of working age. The importance of job retention has been formalized in the objectives of the latest cancer plans, and in the 2018-2022 national health strategy. Initiatives are observed to promote this issue by employers: development of a charter by the National Cancer Institute and in the associative field aimed at promoting support practices in their professional environment for people with cancer. Despite the development of descriptive knowledge on prognostic factors for returning to work after cancer, the results of interventional studies are mixed. No intervention has been shown to be effective in facilitating return to work and reducing social disparities in employment after breast cancer. Interventions have been criticized for being too medicalized and lacking a sufficient theoretical basis to analyse causes (theory of the problem) and propose solutions (theory of action).

The "FASTRACS" intervention was developed with the Intervention Mapping protocol to facilitate the return to work after breast cancer, it defines a return-to-work path from the hospital to the company through care primaries. This intervention is anchored in primary care with an early transition consultation in general medicine in the month following the end of active treatments (chemotherapy or radiotherapy according to the care protocol). This positioning in primary care allows a bio-psycho-social assessment of the needs of women after cancer. This consultation was designed to establish a plan of care and return to work according to the temporality and individual needs of each woman. It will make it possible to determine the right time for the pre-recovery visit in order to anticipate the professional challenges of the recovery.

Return to work/maintenance in employment interventions are complex social interventions, implemented by social actors who act in an environment with which they interact. These interventions (or programs) present an increased risk of failure in their implementation and sustainability. Realistic evaluation comes from the trend of theory-based evaluation (theory-based or theory-driven evaluation). According to this approach, social interventions are based on theories, which can be tested through empirical observation to better understand how and why they produce their effects, and in what context. This approach overcomes the limits of the "black box" model. It is recommended to inform the public decision to interrupt, modify or intensify an intervention. It aims to answer the question: "what works, how, why, for whom, and under what circumstances?" ". It aims to describe the mechanisms of the effectiveness of an intervention by linking its effects to the characteristics of its implementation context (search for CME configurations = context - mechanisms - effects). The search for these configurations, otherwise called "half-regularities" because they can be observed empirically with certain variations, is intended to develop a middle-range theory with a sufficient level of generalization and abstraction. to explain the tendencies and the regularities observed in the interactions contexts-mechanisms-effects of the intervention. This approach is particularly indicated in the evaluation of the FASTRACS intervention, given the complexity of the intervention, the number of actors involved, and the variety of its implementation contexts.

ELIGIBILITY:
* Inclusion Criteria concerning FASTRACS-RCT participants (groupe 1) * :

  * Patients included in the intervention arm of the "FASTRACS-RCT" trial who have completed their participation in the trial.
  * Woman aged between 18 and 55.
  * With a diagnosis of invasive breast carcinoma of stage cTNM or pTNM stage I to III (UICC 8th edition), confirmed on histological examination.
  * Treated by intravenous cytotoxic chemotherapy in an adjuvant or neoadjuvant situation.
  * Breast surgery +/- of the axillary area, carried out within 3 months preceding the start of adjuvant chemotherapy, or scheduled after neoadjuvant chemotherapy +/- radiotherapy.
  * In salaried employment at the time of diagnosis (permanent or temporary contract, interim assignment, civil servant).
  * Affiliated to a French social security scheme.
  * Reading, understanding, and writing the French language.
  * Followed in one of the investigating centers.
  * Not opposing the collection data.
* Inclusion Criteria * :

  * Persons declared by the patients for the study of the trajectories and only if their agreement is obtained for each person concerned (general practitioner, occupational physician, personnel of the resource center fort occupational and environmental pathologies (CRPPE), colleagues and hierarchy in the company and any key person identified by the patient who participated in the recovery process using the intervention tools).(groupe 2)
  * Participants in discussion groups independent of trajectories (oncologists, clinical research associates, general practitioners, occupational health teams and CRPPE staff). (Groupe 3)
  * For all categories of participants, it is necessary to be of legal age, to be able to read, understand and speak French.
* Exclusion Criteria concerning FASTRACS-RCT participants (groupe 1)* :

  * In situ carcinoma.
  * Distant metastases.
  * History or co-existence of another primary cancer (apart from a basal cell cancer of the skin and/or non-mammary cancer in complete remission for more than 5 years).
  * Recurrence or second breast cancer.
  * Without employment contract, self-employed or supported contract.
  * Cannot be followed for the duration of the study, for medical, social, family, geographical or psychological reasons.
  * Deprived of liberty by court or administrative decision.
* Exclusion Criteria * :

  * No exclusion criteria concern participants related to patients (declared by patients) (groupe 2).
  * No exclusion criteria for the people delivering the intervention (focus group participants) (groupe 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients included in the intervention arm of the "FASTRACS-RCT" randomized controlled trial (NCT04846972), the people around them with whom they will have used the FASTRACS intervention tools, their oncologists, the clinical research associates who gave them the intervention documents, their general practitioners, their occupational health service, their colleagues, hierarchies and human resources services within their company and the Resource Center Occupational and Environmental Pathologies (CRPPE) at the Lyon South Hospital Center (HCL).
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Individual semi-directive interviews on barriers and facilitators to the implementation of FASTRACS-RCT intervention | Individual interviews will be conducted from the end of their follow-up in FASTRACS-RCT, and during the following 18 months.
  To identify barriers and facilitators to the implementation of FASTRACS-RCT intervention, we will measure the return-to-work mechanism of women who have had breast cancer, using a 29-question semi-structured interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle de Santé Publique des Hospices Civils de Lyon, Lyon, France